CLINICAL TRIAL: NCT05115370
Title: Barriers and Facilitators of Flu, Pneumonia and SARS-CoV-2 (COVID-19) Vaccination in Adults With Inflammatory Conditions Treated With Immune-suppressing Drugs
Brief Title: Vaccination Perception in Inflammatory Conditions - Flu, Pneumonia and COVID-19
Acronym: OPINION
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 21054
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2021-10

CONDITIONS: Inflammatory Disease; Rheumatoid Arthritis; Psoriatic Arthritis; Systemic Lupus Erythematosus; Ankylosing Spondylitis; Vasculitis; Reactive Arthritis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Lupus Erythematosus, Systemic; Spondylitis, Ankylosing; Vasculitis; Arthritis, Reactive; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with an inflammatory disease taking immune-suppressing medication
  Interventions: Other: Semi-structured qualitative interview

INTERVENTIONS:
Other: Semi-structured qualitative interview — A single semi-structured qualitative interview conducted face-to-face or by telephone or video-conference call.

SUMMARY:
People with inflammatory diseases are often treated with medications that act to suppress the immune-system, increasing the risk of catching infections. Consequently, vaccination with the pneumonia and seasonal flu vaccines is recommended for them. They were also prioritised to receive the COVID-19 vaccines early in the national rollout.

However, the uptake of the pneumonia and seasonal flu vaccines among this group is lower than ideal. There may be many reasons why they do or do not seek to be vaccinated for these infections, such as the belief it may cause their disease to flare up or lack of knowledge of vaccines effectiveness. Anecdotally there was a high uptake of COVID-19 vaccines in adults with inflammatory conditions, however, concerns about vaccine-induced disease flare-ups and reports of complications deterred some from being vaccinated. A better understanding of why people do and do not seek vaccination may result in more targeted messaging for patients to help overcome vaccine hesitancy for these infectious diseases.

This study aims to explore the drivers and barriers to being vaccinated among adults with common inflammatory conditions and on immune-suppressing medication. They will be invited to participate in a single, semi-structured interview. Interviews will be face-to-face, by telephone or video-call, last up to one hour, and digitally audio-recorded. They will explore participants' understanding of pneumonia, seasonal flu and COVID-19 and the risk they pose to their health, their understanding of vaccinations, beliefs of the benefits and risks of vaccinations for these infections, and reasons for seeking or not seeking vaccination.

Findings will inform messaging about being vaccinated for these infections in patient education leaflets, such as those by patient charities regularly provided at speciality clinics. They will also be disseminated to healthcare professionals to help them better understand the drivers and barriers to vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age at-least 18 years,
* Diagnosed with either rheumatoid arthritis, inflammatory bowel disease, psoriatic arthritis, ankylosing spondylitis, systemic lupus erythematosus, vasculitis (small or large vessel), or reactive arthritis, and
* At-least one prescription of either methotrexate, azathioprine, 5-mercaptopurine, sulfasalazine, mycophenolate mofetil, leflunomide, ciclosporin, tacrolimus, or sirolimus, biologic agents (such as anti-TNF, anti-CD 20 etc).
* Ability to give informed consent

Exclusion Criteria:

* Age < 18 years
* Dementia: making it impossible to give informed consent and to comply with interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with an inflammatory condition and on immune-suppressing medication
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Participants' understanding of the flu, pneumonia and Covid-19 respiratory infections and the risks they pose to the health and well-being of people on immune-suppressing treatments | 1 day
  This will be determined through interview
Participants' understanding regarding vaccinations for these infections and how they work | 1 day
  This will be determined through interview
Participants' views about the perceived benefits and risks of vaccination for these infections | 1 day
  This will be determined through interview
The reasons for vaccine uptake versus vaccine hesitancy | 1 day
  This will be determined through interview
The impact of the Covid-19 pandemic on perceptions and engagement with routinely administered vaccinations in this population. | 1 day
  This will be determined through interview

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Abhishek, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided